CLINICAL TRIAL: NCT01091532
Title: A Double Blind, Randomized 3rd Party Open, Placebo Controlled, Parallel Group Multiple Oral Escalating Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of UK-396,082 In Healthy Subjects
Brief Title: A Study In Healthy People Of Multiple Doses Of UK-396,082 Given By Mouth, To Investigate The Safety, Toleration And Time Course Of Blood Concentration Of UK-396,082 And Its Effects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A3941010
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Phase 1; Multiple Dose; Safety; Toleration; Pharmacokinetic
MeSH Terms: interventions — 5-amino-2-((1-n-propyl-1H-imidazol-4-yl)methyl)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Subjects will be assigned to receive either UK-396,082 or placebo
  Interventions: Drug: UK-396,082; Drug: placebo
- Cohort 2 (Experimental): Subjects will be assigned to receive either UK-396,082 or placebo
  Interventions: Drug: UK-396,082; Drug: placebo
- Cohort 3 (Experimental): Subjects will be assigned to receive either UK-396,082 or placebo
  Interventions: Drug: UK-396,082; Drug: placebo
- Cohort 4 (Experimental): Subjects will be assigned to receive either UK-396,082 or placebo
  Interventions: Drug: UK-396,082; Drug: placebo

INTERVENTIONS:
Drug: UK-396,082 — 100mg given orally twice daily for 14 days
  The decision to proceed to the next higher dose will be made jointly by the Pfizer Study Team and the Investigator after careful review of available safety, tolerability and PK information from previous cohorts and dosing periods. The doses will be selected such that the predicted Cmax will not exceed 2.95 mcg/mL and/or the predicted increase in exposure will not exceed 3.5-fold that of the previously studied dose.
  Arms: Cohort 1
Drug: placebo — given orally twice daily for 14 days
  Arms: Cohort 1
Drug: UK-396,082 — 300mg given orally twice daily for 14 days
  The decision to proceed to the next higher dose will be made jointly by the Pfizer Study Team and the Investigator after careful review of available safety, tolerability and PK information from previous cohorts and dosing periods. The doses will be selected such that the predicted Cmax will not exceed 2.95 mcg/mL and/or the predicted increase in exposure will not exceed 3.5-fold that of the previously studied dose.
  Arms: Cohort 2
Drug: placebo — given orally twice daily for 14 days
  Arms: Cohort 2
Drug: UK-396,082 — 1000mg given orally twice daily for 14 days
  The decision to proceed to the next higher dose will be made jointly by the Pfizer Study Team and the Investigator after careful review of available safety, tolerability and PK information from previous cohorts and dosing periods. The doses will be selected such that the predicted Cmax will not exceed 2.95 mcg/mL and/or the predicted increase in exposure will not exceed 3.5-fold that of the previously studied dose.
  Arms: Cohort 3
Drug: placebo — given orally twice daily for 14 days
  Arms: Cohort 3
Drug: UK-396,082 — UK-396,082 given orally, once on Days 1 & 14, and twice daily on Days 3-13.
  The decision to proceed to the next higher dose will be made jointly by the Study Team and the Investigator after careful review of available safety, tolerability and PK information from previous cohorts. Dependent on the emerging safety, tolerability and PK data, Cohort 4 may be recruited to study a higher (or lower) dose of UK-396,082 in order to characterize further the safety, toleration and PK and/or to define the maximum tolerated dose. The dose in Cohort 4 will be selected such that the predicted Cmax will not exceed 46 mcg/mL and/or the predicted increase in exposure will not exceed 3.5-fold that of the previously studied dose.
  Arms: Cohort 4
Drug: placebo — given orally, once on Days 1 & 14, and twice daily on Days 3-13.
  Arms: Cohort 4

SUMMARY:
The purpose of this study in healthy people is to investigate the safety, toleration and time course of UK-396,082 concentration in the blood and any changes in relevant markers of drug effects, following multiple doses given twice daily by mouth for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
safety & toleration: Adverse events, vital signs, 12 lead ECG, blood and urine safety tests and physical examination. | 14 days

SECONDARY OUTCOMES:
Plasma pharmacokinetics: Cmax, Tmax, AUCtau, t½, Rac (=AUCtau (Day 14)/AUCtau (Day 1)), CL/F, Vz/f, Cmin, Cav Urine pharmacokinetics: Aetau & Aetau%, CLR on Day 14 | 14 days
Time course of changes in prothrombin time, activated partial thromboplastin time, TAFi inhibition, fibrinogen and D-dimer concentrations. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3941010&StudyName=A%20Double%20Blind%2C%20Randomized%203rd%20Party%20Open%2C%20Placebo%20Controlled%2C%20Parallel%20Group%20Multiple%20Oral%20Escalating%20Dose%20Study%20to%20Investigate%20the%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20and%20Pharmacodynamics%20of%20UK-396%2C082%20In%20Healthy%20Subjects